CLINICAL TRIAL: NCT00925262
Title: A Controlled Trial of Mental Health Interventions for Common Mental Health Problems Experienced by Torture Survivors Living in Kurdistan, Iraq.
Brief Title: Controlled Trial of Mental Health Interventions for Torture Survivors in Kurdistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Paul Bolton, Associate Scientist, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BoltonP-1
Record Dates: First submitted 2009-06-03; First posted 2009-06-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Depression
Keywords: mental health; randomized controlled trial; torture
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitive Processing Therapy (Experimental): An adaptation of cognitive behavioral therapy, focusing on treatment for persons suffering mental health effects of trauma
  Interventions: Behavioral: Cognitive Processing Therapy
- Behavioral Activation (Experimental): A form of counseling therapy that emphasizes enhancing pleasurable behaviors and minimizing negative behaviors as a means to reducing depression symptomatology.
  Interventions: Behavioral: Behavioral Activation
- non-specific counseling (Experimental): a collection of counseling skills suitable for a broad range of mental health and psychosocial problems and not designed for specific disorders. This particular version was developed by a collaborator -Heartland Alliance - for use with torture survivors.
  Interventions: Behavioral: nonspecific counseling
- wait control (No Intervention): persons in this study arm will not receive active treatment as part of the study but will be monitored during the study and offered treatment after 3-5 months of waiting.

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — an adaptation of cognitive behavioral therapy used to address mental health effects of trauma exposure
  Other Names: CPT
  Arms: Cognitive Processing Therapy
Behavioral: Behavioral Activation — form of counseling intervention to promote positive behaviors and reduce negative behaviors as a means of reducing depression symptomatology and severity
  Other Names: BA
  Arms: Behavioral Activation
Behavioral: nonspecific counseling — nonspecific counseling interventions useful for a broad range of mental health and psychosocial problems.
  Arms: non-specific counseling

SUMMARY:
The purpose of this study is to determine the relative effectiveness of three different mental health counseling interventions in the treatment of mental health problems commonly affecting torture and trauma survivors living in Kurdistan, Iraq.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Kurdish
* torture survivor
* currently has significant depression symptomatology.

Exclusion Criteria:

* danger to self or others
* already receiving treatment from our treatment provider
* not mentally competent to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
depression symptom severity | 3-6 months

SECONDARY OUTCOMES:
ability to carry out routine tasks and activities | 3-6 months
anxiety symptom severity | 3-6 months
posttraumatic stress disorder symptom severity | 3-6 months
traumatic grief symptom severity | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Bolton, MB BS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- multiple public health clinics across Kurdistan, Dohuk, Sulaimani, Erbil, Rural Areas, ALL, Iraq

REFERENCES:
- [Derived] Bolton P, Bass JK, Zangana GA, Kamal T, Murray SM, Kaysen D, Lejuez CW, Lindgren K, Pagoto S, Murray LK, Van Wyk SS, Ahmed AM, Amin NM, Rosenblum M. A randomized controlled trial of mental health interventions for survivors of systematic violence in Kurdistan, Northern Iraq. BMC Psychiatry. 2014 Dec 31;14:360. doi: 10.1186/s12888-014-0360-2. PMID 25551436